CLINICAL TRIAL: NCT01192113
Title: An Open-label, Randomized, Multi-center Clinical Trial to Evaluate the Safety and Efficacy in Peripheral Neuropathies Patients Treated With Mecobalamin Injection
Brief Title: Safety and Efficacy of Mecobalamin Injection in Peripheral Neuropathies Patients (Study JGAZSY091109)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JGAZSY091109
Record Dates: First submitted 2010-08-26; First posted 2010-08-31 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Peripheral Neuropathy
Keywords: Mecobalamin; peripheral neuropathy; diabetic neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Diabetic Neuropathies | interventions — Injections, Intramuscular

ARMS (5):
- Group A: Diabetic Peripheral Neuropathy (IV) (Experimental)
  Interventions: Drug: Mecobalamin IV Injection
- Group B: Diabetic Peripheral Neuropathy (IM) (Experimental)
  Interventions: Drug: Mecobalamin IM injection
- Group C: Idiopathic Peripheral Neuropathy (Experimental)
  Interventions: Drug: Mecobalamin IV or IM injection
- Group D: Nutritional & Metabolic Peripheral Neuropathy (Experimental)
  Interventions: Drug: Mecobalamin IV or IM injection
- Group E: Compression Peripheral Neuropathy (Experimental)
  Interventions: Drug: Mecobalamin IV or IM injection

INTERVENTIONS:
Drug: Mecobalamin IV Injection — Mecobalamin injection 0.5 mg/ ml administered as an intravenous (IV) injection 3 times a week for four weeks
  Arms: Group A: Diabetic Peripheral Neuropathy (IV)
Drug: Mecobalamin IM injection — Mecobalamin injection 0.5 mg/ ml administered as an intramuscular (IM) injection 3 times a week for four weeks
  Arms: Group B: Diabetic Peripheral Neuropathy (IM)
Drug: Mecobalamin IV or IM injection — Mecobalamin injection 0.5 mg/ ml administered as an IM or IV injection 3 times a week for four weeks
  Arms: Group C: Idiopathic Peripheral Neuropathy; Group D: Nutritional & Metabolic Peripheral Neuropathy; Group E: Compression Peripheral Neuropathy

SUMMARY:
This is an open-label, randomized, multi-center clinical trial to evaluate the safety and efficacy in peripheral neuropathies patients treated with Mecobalamin Injection

ELIGIBILITY:
Inclusion criteria:

1. Clinical diagnosis of diabetes induced peripheral neuropathy, other peripheral neuropathies (Idiopathic, nutritional and metabolic nature of entrapment neuropathy).
2. Significant spontaneous pain and / or numbness and other symptoms of neuropathy. TSS (Total Symptom Score) >=7.5.
3. Participation in clinical trials voluntarily and signed informed consent form

Exclusion criteria:

1. Pregnancy, preparation for pregnancy or breast-feeding women
2. Peripheral neuropathy caused by drugs, poisoning, cancer or genetic
3. Alanine aminotransferase (ALT), aspartate aminotransferase (AST): 2.0 times more than the upper limit of normal; Creatinine (Cr) 1.5 times above the upper limit of normal.
4. Serious organ disease or other serious primary disease merger, the mentally ill, poorly controlled hypertension (blood pressure more than 150/100 mmHg after using antihypertensive drugs)
5. Diagnosis of patients with diabetic peripheral neuropathy, but has diabetes ketosis, ketoacidosis and severe infection within the past two weeks
6. Bleeding or bleeding tendency in 2 months
7. Have allergy
8. Noncompliance or cannot meet those
9. Participation in other clinical trials in the last 3 months
10. Participant unsuitable to participate in this test as investigator considering

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1072 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Value of the Peripheral Neuropathy Total Symptom Score (TSS) Compared to Baseline | Baseline & End of Week 4
  The TSS of peripheral neuropathy is used to score the intensity & frequency of four symptoms in participants' feet/legs including: pain, burning sensation, numbness, and hypoesthesia. Frequency is ranked as asymptomatic, occasionally (2-3 times/ week), often (1-2 times/ day), & continuous (nearly all day). Intensity is evaluated by visual analogue scale (VAS) score: 0 (zero intensity)- 10 (max. intensity). Participants described intensity by marking the number corresponding to severity of symptom they felt in a 10 cm long straight line and investigators distinguished whether it was mild (score: 1-3), moderate (score: 4-6), or severe (score: 7-10). The total score of four symptoms was considered the TSS. Total scores ranged from 0-14.64 points, where 0 was lowest symptom score and 14.64 was most severe level of symptoms. Baseline (before treatment) scores were compared to scores after 4 weeks of treatment.
Rate of the Peripheral Neuropathy Total Symptom Score (TSS) Compared to Baseline | Baseline and End of Week 4
  TSS of peripheral neuropathy is used to score the intensity & frequency of 4 symptoms in participants' feet/legs including: pain, burning sensation, numbness, hypoesthesia. Frequency is ranked as asymptomatic, occasionally (2-3 times/ week), often (1-2 times/ day), & continuous (nearly all day). Intensity is evaluated by visual analogue scale (VAS) score: 0 (zero intensity)- 10 (max. intensity). Participants described intensity by marking the number corresponding to severity of symptom they felt in a 10 cm long straight line and investigators distinguished whether it was mild (score: 1-3), moderate (score: 4-6), or severe (score: 7-10). The total score of four symptoms was considered the TSS. Total scores ranged from 0-14.64 points, where 0 was lowest symptom score and 14.64 was most severe level of symptoms. Baseline scores were compared to TSS decreasing rate after 4 weeks of treatment. Rate of TSS change = (TSS difference value/TSS before treatment)×100%.

SECONDARY OUTCOMES:
Value of the Peripheral Neuropathy Total Symptom Score (TSS) Compared to Baseline | Baseline and End of Week 2
  The TSS of peripheral neuropathy is used to score the intensity & frequency of four symptoms in participants' feet/legs including: pain, burning sensation, numbness, and hypoesthesia. Frequency is ranked as asymptomatic, occasionally (2-3 times/ week), often (1-2 times/ day), & continuous (nearly all day). Intensity is evaluated by visual analogue scale (VAS) score: 0 (zero intensity)- 10 (max. intensity). Participants described intensity by marking the number corresponding to severity of symptom they felt in a 10 cm long straight line and investigators distinguished whether it was mild (score: 1-3), moderate (score: 4-6), or severe (score: 7-10). The total score of four symptoms was considered the TSS. Total scores ranged from 0-14.64 points, where 0 was lowest symptom score and 14.64 was most severe level of symptoms. Baseline (before treatment) scores were compared to scores after 2 weeks of treatment.
Rate of the Peripheral Neuropathy Total Symptom Score (TSS) Compared to Baseline | Baseline and End of Week 2
  TSS of peripheral neuropathy is used to score the intensity/ frequency of 4 symptoms in participants' feet/legs including: pain, burning sensation, numbness, and hypoesthesia. Frequency is ranked as asymptomatic, occasionally (2-3 times/ week), often (1-2 times/ day), & continuous (nearly all day). Intensity is evaluated by visual analogue scale (VAS) score: 0 (zero intensity)- 10 (max. intensity). Participants described intensity by marking the number corresponding to severity of symptom they felt in a 10 cm long straight line and investigators distinguished whether it was mild (score: 1-3), moderate (score: 4-6), or severe (score: 7-10). The total score of four symptoms was considered the TSS. Total scores ranged from 0-14.64 points, where 0 was lowest symptom score and 14.64 was most severe level of symptoms. Baseline scores were compared to TSS decreasing rate after 2 weeks of treatment. Rate of TSS change = (TSS difference value/TSS before treatment)×100%.
Value of the Neural Injury Score of the Lower Limbs (NIS-LL) Compared to Baseline | Baseline and End of Week 4
  The Neural Injury Score of the Lower Limbs (NIS-LL) was scored based on the following examination items: muscle strength (including hip & knee flexion/ extension & remote foot dorsiflexion/ plantar flexion [scored as normal, 25% weak, 50% weak, 75% weak, and paralysis]), reflex (response at the quadriceps & ankle [normal score=0, decreased score=1, absent score=2], and sensory (tested at the great toe; including touch pressure, pinprick ,vibration, and joint position [normal score=0, decreased score=1, absent score=2]). The Total NIS-LL score ranged from 0-8 points where a higher score means greater neural injury of the lower limbs. Baseline (before treatment) scores were compared to scores after 4 weeks of treatment.
Rate of the Neural Injury Score of the Lower Limbs (NIS-LL) Compared to Baseline | Baseline and End of Week 4
  The Neural Injury Score of the Lower Limbs (NIS-LL) was scored based on the following examination items: muscle strength (including hip & knee flexion/ extension & remote foot dorsiflexion/ plantar flexion [scored as normal, 25% weak, 50% weak, 75% weak, and paralysis]), reflex (response at the quadriceps & ankle [normal score=0, decreased score=1, absent score=2], and sensory (tested at the great toe; including touch pressure, pinprick ,vibration, and joint position [normal score=0, decreased score=1, absent score=2]). The Total NIS-LL score ranged from 0-8 points where a higher score means greater neural injury of the lower limbs. Baseline (before treatment) scores were compared to scores after 4 weeks of treatment. Rate of NIS-LL change = (NIS-LL difference value/NIS-LL before treatment)×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Jvming Lu, Principal Investigator — Chinese PLA General Hospital
Locations (24):
- China (24):
  - The 1st Hospital of Anhui Medical University, Hefei, Anhui
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - The institute of rehabilitation medicine, Beijing, Beijing Municipality
  - Nanfang Hospital of Nanfang Medical Unversity, Guangzhou, Guangdong
  - The 1st People Hospital of Guangzhou, Guangzhou, Guangdong
  - the 1st Hospital affliated to Guangxi Medical University, Nanning, Guangxi
  - The 3rd Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - the people Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Xiehe Hospital, Wuhan, Hubei
  - the 1st Hospital of Nanjing, Nanjing, Jiangsu
  - Zhong Xi Yi Jie He Hospital of Jiangsu, Nanjing, Jiangsu
  - the 2nd Hospital of Suzhou University, Suzhou, Jiangsu
  - Subei People Hospital, Yangzhou, Jiangsu
  - The 1st People Hospital of Yangzhou, Yangzhou, Jiangsu
  - the Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Ruijing Hospital, Shanghai, Shanghai Municipality
  - the 10th People Hospital of Shanghai, Shanghai, Shanghai Municipality
  - the 10th People Hospital, Shanghai, Shanghai Municipality
  - The 1st Center Hospital of Tianjin, Tianjin, Tianjin Municipality
  - The institute of rehabilitation medicine, Beijing
  - Rui Jin Hospital, Shanghai
  - Shenzhen Hospital of Beijing University, Shenzhen